CLINICAL TRIAL: NCT07179575
Title: Phase Ib/II Study of LW231 in Patients With Chronic Hepatitis B: Evaluation of Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy With Multiple-Dose, Dose-Escalation, and Combination With Nucleos(t)Ide Analogs (NUC)
Brief Title: Study of LW231 in Participants With Chronic Hepatitis B
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Longwood Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LW231-Ib/II-01
Record Dates: First submitted 2025-09-16; First posted 2025-09-18 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Chronic HBV Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part1: LW231 Dose 1 (Experimental): LW231 Dose Escalation Cohort 1, administered orally, QD
  Interventions: Drug: LW231; Drug: LW231 placebo
- Part1: LW231 Dose 2 (Experimental): LW231 Dose Escalation Cohort 2, administered orally, BID
  Interventions: Drug: LW231; Drug: LW231 placebo
- Part1: LW231 Dose 3 (Experimental): LW231 Dose Escalation Cohort 2, administered orally, QD
  Interventions: Drug: LW231; Drug: LW231 placebo
- Part2: LW231 treatment group 1 (Experimental): LW231 administered orally, BID + NUCs
  Interventions: Drug: LW231
- Part2: LW231 treatment group 2 (Experimental): LW231 administered orally, QD +NUCs
  Interventions: Drug: LW231
- Part2: LW231 placebo group (Placebo Comparator): LW231 placebo + NUCs
  Interventions: Drug: LW231 placebo

INTERVENTIONS:
Drug: LW231 — LW231 tablets
  Arms: Part1: LW231 Dose 1; Part1: LW231 Dose 2; Part1: LW231 Dose 3; Part2: LW231 treatment group 1; Part2: LW231 treatment group 2
Drug: LW231 placebo — LW231 placebo tablets
  Arms: Part1: LW231 Dose 1; Part1: LW231 Dose 2; Part1: LW231 Dose 3; Part2: LW231 placebo group

SUMMARY:
This is a Phase Ib/II, multicenter, randomized, dose-escalation study designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of LW231 in participants with chronic hepatitis B virus (HBV) infection. The trial will include multiple-dose regimens of LW231 and assess LW231 in combination with NUCs.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: treatment-naïve and currently not treated subjects: LLOQ<HBV DNA≤20000 IU/ml; 100 IU/mL<HBsAg<10000 IU/ml
* Part 2: HBV DNA<LLOQ or < 20 IU/mL at screening; 100 IU/mL<HBsAg<3000 IU/mL

Exclusion Criteria:

* Co-infection with hepatitis A, C, D, E or HIV or any evidence of clinically significant liver disease of non-HBV etiology.
* History or current evidence of cirrhosis.
* ALT or AST>3×ULN; TBil>1.3×ULN or DBil>1.3×ULN; INR>1.3×ULN

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in HBV DNA Viral Load Assay | 4 weeks

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | up to 28 weeks
  An adverse event (AE) was defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product (including investigational drug) during the course of a clinical investigation. An AE could therefore be any unfavorable and unintended sign (including abnormal laboratory findings), symptom, or disease that was temporally associated with the use of the investigational product, regardless of whether it was considered to be related to the investigational product or not.
Change from baseline in HBsAg | Up to 28 weeks
Maximum Plasma Concentration (Cmax) of LW231 | Up to 28 Weeks
Area Under the Curve From Time 0 to the Last Measurable Concentration (AUClast) of LW231 | Up to 28 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou

IPD SHARING:
Plan to Share IPD: No